CLINICAL TRIAL: NCT03604484
Title: Prophylactic Tricuspid Annuloplasty During Mitral Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Pettinari Matteo, Principal Investigator, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCLSaint Luc
Record Dates: First submitted 2018-07-11; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Tricuspid Valve Insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tricuspid annuloplasty (Active Comparator): Patient treated with tricuspid annuloplasty at the moment of the mitral valve surgery
  Interventions: Procedure: Tricuspid annuloplasty
- No Tricuspid annuloplasty (No Intervention): Control patients

INTERVENTIONS:
Procedure: Tricuspid annuloplasty — Tricuspid annuloplasty
  Arms: Tricuspid annuloplasty

SUMMARY:
Single center randomized study to test whether a prophylactic tricuspid annuloplasty at the time of mitral valve procedure can improve clinical and echocardiographical outcomes.

DETAILED DESCRIPTION:
The optimal management of functional tricuspid regurgitation (FTR) in the setting of mitral valve operations remains controversial. The current practice is both center- and surgeon-specific with guidelines based on non-randomized data. A prospective randomized trial was performed to evaluate the worth of less-than-severe FTR repair during mitral valve procedures.

A single center randomized study was designed to allocate patients with less-than-severe FTR undergoing mitral valve surgery to be prophylactically treated + tricuspid valve annuloplasty (TVP- or TVP+). These patients were analysed using longitudinal cardiopulmonary exercise capacity, echocardiographic follow-up, and cardiac magnetic resonance (CMR). The primary outcome was more than mild tricuspid regurgitation (TR) recurrence with vena contracta >3mm. Secondary outcomes were maximal oxygen uptake (VO2 max) and right ventricular (RV) dimension and function.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing mitral valve surgery with less than sever tricuspid insufficiency

Exclusion Criteria:

* presence of pacemaker lead through the tricuspid valve
* acute endocarditis
* minimally invasive approach
* Functional mitral valve insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of more than mild tricuspid insufficiency | 5 year

SECONDARY OUTCOMES:
VO2 max | 1 year
  Physical function capacity measured by VO2 max
Right ventricular function | 5 year
  Right ventricle function at the follow up